CLINICAL TRIAL: NCT04707573
Title: A Phase 2A Single Dose, Open Label Study to Assess the Safety and Pharmacokinetics of AKB-6548 in Subjects With Chronic Kidney Disease (CKD), Stages 3 and 4
Brief Title: Study to Assess the Safety and Pharmacokinetics of AKB-6548 in Participants With Chronic Kidney Disease (CKD), Stages 3 and 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0003
Record Dates: First submitted 2020-11-02; First posted 2021-01-13 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Chronic Kidney Disease
Keywords: CKD; CKD, Stage 3; CKD, Stage 4; Vadadustat; pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — vadadustat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CKD, Stage 3 (Experimental): Participants with Stage 3 Chronic Kidney Disease (CKD) (Estimated Glomerular Filtration Rate [eGFR] 30 - 59 milliliters [mL]/minute) received a single 500 milligram (mg) oral dose of Vadadustat after fasting for at least 4 hours.
  Interventions: Drug: Vadadustat
- CKD, Stage 4 (Experimental): Participants with Stage 4 CKD (eGFR <30 mL/minute and not yet on dialysis) received a single 500 mg oral dose of Vadadustat after fasting for at least 4 hours.
  Interventions: Drug: Vadadustat

INTERVENTIONS:
Drug: Vadadustat — oral capsules
  Other Names: AKB-6548

SUMMARY:
This study was conducted to assess the pharmacokinetic (PK) profile, safety, and tolerability in participants with Stage 3 and 4 Chronic Kidney Disease (CKD) following a single oral dose of Vadadustat.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 79 years of age, inclusive
* Chronic Kidney Disease Stage 3 (Estimated Glomerular Filtration Rate [eGFR] 30 to 59 milliliters [mL]/minute) or Stage 4 participants (eGFR of <30 mL/minute that were not yet on dialysis). eGFR was calculated using the Modification of Diet in Renal Disease (MDRD).
* Hemoglobin (Hb) <13.5 grams per deciliter (g/dL) except for Polycystic Kidney Disease (PKD) participants, in which Hb was to be ≤14 g/dL
* Transferrin saturation (TSAT) >12% and complete blood count (CBC) indicating normocytic red blood cell morphology, unless the medical monitor and investigator agreed that the participant was appropriate for this study
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤1.8 x upper limit of normal (ULN)
* Alkaline phosphatase ≤2 x ULN
* Bilirubin ≤1.5 x ULN
* Female participants were not pregnant or breastfeeding. Women of childbearing potential agreed to use an acceptable method of contraception.
* Non-vasectomized male participants agreed to use an acceptable method of contraception
* Understood the procedures and requirements of the study and provided written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Any medical or psychological condition that in the opinion of the Investigator would have interfered with the participant's ability to provide informed consent or comply with study instructions
* Any clinically significant or uncontrolled medical condition that in the opinion of the Investigator would have placed the participant at undo risk or would have compromised the interpretability of the findings in this study
* A body mass index (BMI) of greater than 40
* Seropositive for human immunodeficiency virus (HIV) or Hepatitis B surface antigen
* Seropositive for Hepatitis C virus (HCV) antibodies unless ALT, AST, bilirubin tests were within normal limits
* History of chronic liver disease
* Uncontrolled hypertension (diastolic blood pressure [BP] > 110 millimeters of mercury [mm Hg] or systolic BP >190 mm Hg at screening)
* New York Heart Association Class III or IV congestive heart failure
* Myocardial infarction, acute coronary syndrome, or stroke within 6 months of dosing
* History of myelodysplastic syndrome
* Participants known to have diabetic gastroparesis that was either symptomatic on therapy or was refractory to therapy
* Any history of malignancy in the previous 5 years except for curatively resected basal cell carcinoma of skin, squamous cell carcinoma of skin, cervical carcinoma in situ, or resected benign colonic polyps
* Evidence of active infection unless the medical monitor and investigator agreed that the participant was appropriate for this study
* History of rheumatoid arthritis or systemic lupus erythematosus (SLE) (History of osteoarthritis or gout did not exclude participants from eligibility in the study.)
* Age-related macular degeneration (AMD), diabetic macular edema or active diabetic proliferative retinopathy that was likely to require treatment during the trial
* History of deep vein thrombosis (DVT) that required active treatment. Superficial thrombosis was not excluded.
* History of ongoing hemolysis or diagnosis of hemolytic syndrome
* Known history of bone marrow fibrosis
* History of hemosiderosis or hemochromatosis
* Androgen therapy within 21 days from the last injection
* Red blood cell transfusion within 12 weeks
* Therapy with an erythropoiesis stimulating agent (ESA) such as human recombinant erythropoietin within the past 21 days
* Intravenous iron supplementation within the past 21 days
* Currently taking acetaminophen > 2.6 grams/day
* History of prior organ transplantation, or stem cell or bone marrow transplantation
* Alcohol consumption greater than 14 or more drinks per week within the past year (1 drink = 12 ounce [oz] beer, 5 oz wine, or 1.5 oz hard liquor.)
* Use of an investigational medication or participation in an investigational study within 30 days, or 5 half-lives of the investigational product, whichever was longer, preceding Day 1
* Positive urine toxicology screen for a substance of abuse that had not been prescribed for the participant

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-07-08 (Actual); Primary Completion 2010-09-24 (Actual); Study Completion 2010-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (2):
- United States (2):
  - Research Site, Saint Paul, Minnesota
  - Research Site, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 22 participants were enrolled in this study. The participants were placed in one of two cohorts, depending on disease state: Chronic Kidney Disease (CKD) Stage 3 (Cohort 1) or CKD Stage 4 (Cohort 2).
Groups:
- Cohort 1: CKD Stage 3 Vadadustat: Participants with CKD Stage 3 with Estimated Glomerular Filtration Rate (eGFR) 30 - 59 milliliter (mL)/minute received a single dose of Vadadustat 500 milligrams (mg) (one 200 mg capsule and one 300 mg capsule) orally in fasted condition.
- Cohort 2: CKD Stage 4 Vadadustat: Participants with CKD Stage 4 with eGFR <30 mL/minute and not yet on dialysis received a single dose of Vadadustat 500 milligrams (mg) (one 200 mg capsule and one 300 mg capsule) orally in fasted condition.
Period: Overall Study
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Population: The enrolled population consisted of all participants who were enrolled in the study.
Groups:
- Cohort 1: CKD Stage 3 Vadadustat: Participants with CKD Stage 3 with Estimated Glomerular Filtration Rate (eGFR) 30 - 59 mL/minute received a single dose of Vadadustat 500 milligrams (mg) (one 200 mg capsule and one 300 mg capsule) orally in fasted condition.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (12.9) | 64.4 (10.0) | 63.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 12 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: mL/min/1.73m^2] — eGFR in normal range (60-89 milliliter/minute/1.73 meter square [mL/min/1.73m^2]) with other signs of kidney damage, like protein in urine or physical damage to the kidneys. eGFR 30-59, moderate kidney damage. eGFR 15-29, severe kidney damage. eGFR less than 15, the kidneys are close to failure or have already failed.
  mL/min/1.73m^2 | 45.22 (8.54) | 24.39 (3.31) | 33.86 (12.23)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was defined as any untoward, undesired, unplanned clinical event in the form of signs, symptoms, disease, or laboratory or physiological observations occurring in a human being participating in a clinical study following study medication administration, regardless of causal relationship. This also included any clinically significant worsening or re-occurrence of a pre-existing condition, or AE occurring from an overdose of a study drug whether accidental or intentional or AE occurring from abuse of study drug or that has been associated with the discontinuation of the use of study drug.
Time Frame: Up to Day 8
Population: Intent-to-treat (ITT) population: all enrolled participants who received a dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Participants | 6 | 2

2. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameter Values
Description: Parameters assessed for laboratory values included hematology, chemistry, urinalysis, and coagulation. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to Day 8
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Participants
  Urinalysis | 0 | 0
  Hematology | 0 | 0
  Serum chemistry | 1 | 0
  Coagulation | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Sign Values
Description: Parameters assessed for vital signs included sitting (at rest for a minimum of 5 minutes) heart rate, respiratory rate, body temperature, and blood pressure. The investigator was responsible for reviewing laboratory results for clinically significant changes. Number of participants with a clinically significant change from baseline in at least one of the assessed vital signs parameters is reported.
Time Frame: Up to Day 8
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Participants | 2 | 0

4. Primary Outcome: Number of Participants With Clinically Abnormal 12-Lead Electrocardiogram (ECG) Findings
Description: A standard 12-lead ECG was performed following dosing in a supine position for approximately 10 minutes. ECGs were taken prior to blood draws when possible. The investigator was responsible for reviewing laboratory results for clinical significance.
Time Frame: Up to Day 2
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

5. Primary Outcome: Change From Baseline in PR Interval, QT Interval, QRS Interval, and QT Corrected (QTc) Interval
Description: A standard 12-lead ECG was performed following dosing in a supine position for approximately 10 minutes. ECGs were taken prior to blood draws when possible. The parameters evaluated from the participant ECG trace included PR interval, QT interval, QRS interval, and QTc (corrected). The baseline was defined as Day 1 pre-dose measurement. If missing, the last measurement prior to dosing was used.
Time Frame: Baseline; Day 2
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Milliseconds
  Baseline PR interval | 178.8 (44.2) | 182.5 (24.2)
  Change from Baseline at Day 2 PR interval | -12.4 (28.4) | -3.5 (5.5)
  Baseline QRS interval | 98.8 (20.7) | 97.7 (26.0)
  Change from Baseline at Day 2 QRS interval | -0.8 (3.2) | 0.0 (5.4)
  Baseline QT interval | 427.2 (22.0) | 426.5 (39.7)
  Change from Baseline at Day 2 QT interval | -13.8 (21.8) | -2.3 (16.7)
  Baseline QTc interval | 423.5 (22.8) | 439.5 (35.8)
  Change from Baseline at Day 2 QTc interval | 3.1 (10.2) | 2.0 (18.2)

6. Primary Outcome: Change From Baseline in Heart Rate
Description: The heart rate evaluation was performed after the participant had been resting comfortably in a supine position for approximately 10 minutes.
Time Frame: Baseline; Day 2
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Beats per minute
  Baseline | 59.8 (9.0) | 64.3 (5.6)
  Change from Baseline at Day 2 | 5.2 (6.3) | 1.8 (3.7)

7. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Physical Examination Findings
Description: A baseline physical examination was performed at screening. Otherwise, abbreviated physical examinations were conducted and were to include heart, lung, and abdomen. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to Day 8
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Participants | 0 | 0

8. Primary Outcome: Geometric Mean Maximum Observed Plasma Concentration (Cmax) of AKB-6548
Description: Plasma samples were collected from the participants at the defined time points. Cmax was defined as the maximum observed plasma concentration. Cmax was calculated using the standard non-compartmental method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose (Day 2)
Population: Pharmacokinetic (PK) Evaluable Population: all ITT participants who had adequate and reliable PK data for the evaluation of PK of AKB-6548 plasma concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per millilitre (mcg/mL)
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Micrograms per millilitre (mcg/mL) | 42.486 (36.314) | 40.952 (35.022)

9. Primary Outcome: Median Time to Reach Cmax (Tmax) of AKB-6548
Description: Plasma samples were collected from the participants at the defined time points. Tmax was defined as the time to reach maximum plasma concentration. Tmax was calculated using the standard non-compartmental method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose (Day 2)
Population: PK Evaluable Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Hours | 5.5 [1.0 to 8.0] | 5.0 [2.0 to 6.0]

10. Primary Outcome: Mean Terminal Elimination Rate Constant (λz)
Description: Plasma samples were collected from the participants at the defined time points. λz was calculated using linear regression of the terminal linear portion of the log concentration vs. time curve. The parameter was calculated by linear least-squares regression analysis using three or more concentrations, excluding Cmax.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose (Day 2)
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: 1/Hour
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
1/Hour | 0.105 (0.029) | 0.086 (0.020)

11. Primary Outcome: Median Terminal Elimination Half-life (T½)
Description: Plasma samples were collected from the participants at the defined time points. T½ was defined as apparent terminal elimination half-life. T½ was calculated using the standard non-compartmental method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose (Day 2)
Population: PK Evaluable Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Hours | 7.070 [4.530 to 9.930] | 7.530 [5.680 to 12.270]

12. Primary Outcome: Geometric Mean Area Under the Plasma Concentration-time Curve From 0 to Time T Over a Dosing Interval (AUC[0-T])
Description: Plasma samples were collected from the participants at the defined time points. AUC[0-T) was defined as the area under the plasma concentration-time curve, from time=0 to the last measurable concentration (Ct) up to 24 hours, calculated by the linear trapezoidal method. AUC[0-T) was calculated using the standard noncompartmental method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose (Day 2)
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
mcg*hr/mL | 441.651 (36.162) | 448.399 (34.081)

13. Primary Outcome: Geometric Mean Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC[0-∞])
Description: Plasma samples were collected from the participants at the defined time points. AUC[0-∞] was defined as the area under the plasma concentration-time curve from time=0 and extrapolated to infinity. AUC[0-∞] was calculated using the standard non-compartmental method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose (Day 2)
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
mcg*hr/mL | 503.688 (41.671) | 535.813 (40.320)

14. Primary Outcome: Geometric Mean Apparent Oral Clearance (CL/F)
Description: Plasma samples were collected from the participants at the defined time points. CL/F was defined as apparent oral clearance, calculated as Dose/AUC(0-inf). CL/F was calculated using the standard non-compartmental method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose (Day 2)
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre per Hour (L/hr)
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Litre per Hour (L/hr) | 0.995 (41.683) | 0.934 (40.324)

15. Primary Outcome: Geometric Mean Apparent Volume of Distribution During the Terminal Phase (Vd/F)
Description: Plasma samples were collected from the participants at the defined time points. Vd/F was defined as the apparent volume of distribution during the terminal phase, calculated as Dose/[λz * AUC(0-inf)]. Vd/F was calculated using the standard non-compartmental method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose (Day 2)
Population: PK Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
Liter | 9.863 (20.479) | 11.105 (31.747)

16. Secondary Outcome: Change From Baseline in Mean Erythropoietin (EPO)
Description: The change from baseline was calculated by subtracting the baseline value from the individual post-dose visit values.
Time Frame: Baseline; 8, 12, and 24 hours post-dose
Population: ITT Population. Overall number of participants analyzed represents participants with valid EPO measurements at both baseline and the post-dose hour.
Measure: Mean (Standard Deviation); unit: milli-international units per milliliter
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
Number analyzed (Participants) | 10 | 12
milli-international units per milliliter
  Baseline | 23.14 (15.00) | 21.65 (15.84)
  8 Hours Post-dose | 6.16 (9.97) | 12.07 (11.13)
  12 Hours Post-dose | 5.41 (7.66) | 11.09 (8.71)
  24 Hours Post-dose | -1.44 (5.71) | 2.08 (5.57)

17. Other Pre Specified Outcome: Exploratory: Change From Baseline in Hepcidin at 24 Hours
Time Frame: Baseline; 24 hours post-dose
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Exploratory: Change From Baseline in Vascular Endothelial Growth Factor (VEGF) at 24 Hours
Time Frame: Baseline; 24 hours post-dose
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Exploratory: Change From Baseline in Transferrin at 24 Hours
Time Frame: Baseline; 24 hours post-dose
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Exploratory: Change From Baseline in Cystatin-C at 24 Hours
Time Frame: Baseline; 24 hours post -dose
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Exploratory: Change From Baseline in Adiponectin at 24 Hours
Time Frame: Baseline; 24 hours post -dose
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Exploratory: Change From Baseline in Ferritin at 24 Hours
Time Frame: Baseline; 24 hours post-dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to Day 8
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, were reported.
Arm/Group | Cohort 1: CKD Stage 3 Vadadustat | Cohort 2: CKD Stage 4 Vadadustat
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 6/10 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: CKD Stage 3 Vadadustat (N=10) | Cohort 2: CKD Stage 4 Vadadustat (N=12)
Tachycardia (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Catheter Site Inflammation (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other